CLINICAL TRIAL: NCT06449872
Title: ECHO-007 OB-GYN Clinical Validation Study
Brief Title: OB-GYN Clinical Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EchoNous Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHO-007
Record Dates: First submitted 2024-05-20; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Obstetric Complication; GYN Disorders
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Comparison scanning protocol for OB and GYN clinical applications (Other): Image quality comparative assessment
  Interventions: Device: Obstetrics and Gynecology clinical applications for ultrasound diagnostic systems

INTERVENTIONS:
Device: Obstetrics and Gynecology clinical applications for ultrasound diagnostic systems — Up to 5 healthcare professionals trained and experienced in Obstetrics and Gynaecology ultrasound qualitatively assessed the diagnostic image quality of the Kosmos Diagnostic Ultrasound System against the benchmark Mindray M9 Ultrasound System.

SUMMARY:
This is a single-site study evaluating obstetrics and gynecology exam imaging quality by expert users.

DETAILED DESCRIPTION:
Six healthcare professionals with training and experience in Obstetrics and Gynecology ultrasound qualitatively assessed the image quality of the Kosmos Diagnostic Ultrasound System compared to the benchmark Mindray M9 Ultrasound System. Five sonographers were required to complete each scanning cohort of at least three gravid and three non-gravid participants. A sixth sonographer was added to the study to accommodate a scheduling conflict and provided additional image quality data outside of the five completed cohorts.

The following views/structures were assessed for image quality:

Gynecology participants:

* Uterus
* Ovaries
* Endometrial cavity
* Cervix

  • Obstetrics participants in their 1st trimester:
* General image quality of the fetus
* Ability to visualize the crown rump length
* Visualization of gestational sac
* Visualization of yolk sac if present

  • Obstetrics and participants in their 2nd trimester:
* General image quality of the fetal structures
* Visualization of the amniotic fluid
* Visualization of the placenta
* Cardiac motion in 2D and M-mode with heart rate

Obstetrics and participants in their 3rd trimester:

* General image quality of the fetal structures
* Visualization of the amniotic fluid
* Visualization of the placenta
* Visualization of the maternal cervix
* Cardiac motion in 2D and M-mode with heart rate
* 3 vessel umbilical cord in 2D and Color Doppler The sonographers captured all views/structures on the Mindray M9 Ultrasound System, then switched over to the Kosmos Diagnostic Ultrasound System to capture the same views/structures. Once all views/structures were captured on both ultrasound systems, the healthcare professionals reviewed the images in parallel on each system, then provided a comparison score for Kosmos between 1 and 7.

ELIGIBILITY:
Inclusion Criteria:

1. Persons able to:

   1. Read and sign an English consent form.
   2. Read and complete an English demographic and general health survey.
   3. Give consent for participation.
   4. Able and willing to comply with study requirements.
2. Those aged 18 years through 40 years, healthy, particularly in respect to their pregnancy.
3. Pregnant individuals who have received a previous ultrasound exam by their physician.

Exclusion Criteria:

1. Children (minors) under 18 years old.
2. Adults over 40 years old.
3. Those who cannot or refuse to sign their consent.
4. Those who cannot provide informed consent.
5. Vulnerable populations, i.e., individuals whose willingness to participate in the study could be unduly influenced by the expectation of medical benefits associated with participation.
6. Vulnerable populations, i.e., individuals whose willingness to participate in the study could be unduly influenced by parents, employer or monetary benefit.
7. Pregnant individuals who have not received a previous ultrasound exam by their physician.
8. Individuals who have had a hysterectomy, oophorectomy, and trachelectomy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Average Ultrasound Image Quality Score | Through study completion, up to 1 month
  Qualitative image assessment of required views/structures generated with Kosmos Diagnostic Ultrasound System versus a cart-based ultrasound system.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Blankenship, MD, Principal Investigator — Mercy West Hospital
Locations (1):
- EchoNous, Inc., Redmond, Washington, United States